CLINICAL TRIAL: NCT05434065
Title: Effects and Mechanisms of Celecoxib on Intracerebral Hemorrhage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202112193MINB
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral hemorrhage; Celecoxib; COX-2 inhibitor
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: Intracerebral hemorrhage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celebrex treatment arm (Experimental): Celecoxib 200 mg/dose, started within 6 h after onset, then one dose per day for 21 days.
  Interventions: Drug: Celecoxib 200mg
- Control arm (No Intervention): No trial medication will be given.

INTERVENTIONS:
Drug: Celecoxib 200mg — Using celecoxib (200 mg/day) for 21 days starting within 6 hours after onset of ICH
  Arms: Celebrex treatment arm

SUMMARY:
This trial is a phase IIa human clinical study, in which 60 patients with intracerebral hemorrhage (ICH) at basal ganglion or thalamus within 6 h after onset will be enrolled. Patients will be randomly assigned as treatment group or control group as 1:1 distribution. Early initiation of celecoxib within 6 h after ICH and treatment for 21 days will be performed. The safety will be evaluated by drug adverse effects. The efficacy will be assessed by hematoma expansion, brain edema, and 3-month modified Rankin scale.

DETAILED DESCRIPTION:
A phase IIa human clinical trial will be performed to clarify the safety and efficacy of using usual dose of celecoxib (200 mg/day) for 21 days starting within 6 hours after onset of ICH. Totally 60 patients will be enrolled prospectively, and the case number was estimated by statistical methods for the percentage of participants with increased perihematomal edema volume shown in the previous clinical trial (Lee et al., 2013) (estimated by G-power software, settings as: exact test, one sample test, α = 0.05, power = 0.95). Patients will be randomly assigned as treatment group or control group as 1:1 distribution.

Intervention: Celecoxib 200 mg per dose, started within 6 h after onset, then one dose per day for 21 days in the treatment group. The low dose of Celecoxib will be used to minimize the side effect of Celecoxib. No trial medication will be given for the control group. Pregnancy will be excluded at enrollment and prevented throughout the treatment period in female cases at reproductive ages.

Evaluations:

1. Brain CT:

   1. Initial brain CT: for initial hematoma volume (length * width * height /2)
   2. Brain CT on day 2 for final hematoma volume and hematoma expansion
   3. Brain CT on day 7±1 for perihematomal edema and hematoma resolution
2. Neurological functions: NIHSS score, GCS score, modified Rankin scale (mRS) on day 1, 2, 7±2, 14±2, 21±2, and mRS at 3 months
3. Renal function (creatinine) on day 1, then once per week during day 2-7, day 8-14 and 15-21
4. Gastrointestinal bleeding evens within 21 days
5. Myocardial infarction evens within 21 days
6. Blood sampling on day 1, 7±2, and 21±2

Patient enrollment: If the patient's consciousness is not clear before the enrollment of this study, his (her) family can decide the enrollment for this patient. Once the patient regains his (her) consciousness, we will reconfirm with the patient about the enrollment of this study.

Data checks: The data recorded of this study will be double-checked for their accuracy and compared with predefined ranges to avoid typing error.

Plan for missing data: Missing data include those data which are reported as missing, unavailable, uninterpretable, or considered missing because of data inconsistency or out-of-range results. This study will try to minimize missing data by limiting the collection of data to essential information and minimizing the number of follow-up visits, develop a documentation of this study for the methods to screen the participants and the procedures to follow up, appropriate training for all personnel related to this study, and data will be reviewed as close to real-time as possible.

Statistical analysis plan: The continuous variables between Celecoxib group and control group will be compared using Mann-Whitney U test if these data are not with normal distribution, or t-test if these data are with normal distribution. Categorical data will be compared using Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* Acute ICH patients able to take the first dose within 6 hours after onset
* ICH location at basal ganglion or thalamus
* ICH volume < 30 mL
* Normal renal function (creatinine [Cr] ≤ 1.3 mg/dL)
* No surgical indication
* Signed informed consent
* Consciousness clear or mild drowsiness
* Age 20-80 years old

Exclusion Criteria:

* Allergy to celecoxib or other non-steroid anti-inflammatory drugs (NSAIDs)
* Post-coronary artery bypass graft (CABG) within 14 days
* Previous myocardial infarction
* Previous peptic ulcer disease
* Abnormal renal function (Cr > 1.3 mg/dL)
* Surgery for this ICH
* Pregnancy or under breast feeding (If the female case is not sure about pregnancy, pregnancy test will be performed)
* Premorbid mRS > or = 3
* Previous ICH not at basal ganglia or thalamus
* Coagulation abnormality (abnormal PT/PTT), or taking anticoagulant or antiplatelet
* Abnormal liver function (ALT > 3x upper limit)
* History of severe bleeding event, requiring admission or blood transfusion
* History of stenting or valve replacement, requiring long-term using antithrombotics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematoma expansion volume percentage | Day 2
  (Followed hematoma volume - initial hematoma volume) / initial hematoma volume x100%
Perihematomal edema change volume percentage | Day 2, 7
  (Followed perihematomal edema volume - initial perihematomal edema volume) / initial perihematomal edema volume x100%
Percentage of participants with perihematomal edema volume change > 20% | Day 2, 7
  Participants with [(followed perihematomal edema volume - initial perihematomal edema volume) / initial perihematomal edema volume x100%] larger than 20% / total participants x100%

SECONDARY OUTCOMES:
Hematoma expansion volume | Day 2
  Followed hematoma volume - initial hematoma volume
Percentage of participants with hematoma expansion (33% relative or 12.5 mL absolute volume increase) | Day 2
  Participants with hematoma expansion on followed CT (33% relative volume increase or 12.5 mL absolute volume increase) / total participants X100%
Perihematomal edema increase volume | Day 2, 7±1
  Followed perihematomal edema volume - initial perihematomal edema volume
Hematoma and perihematomal edema expansion volume | Day 2, 7±1
  Total volume of hematoma and perihematomal edema on followed CT - initial total volume of hematoma and perihematomal edema
Hematoma and perihematomal edema expansion percentage | Day 2, 7±1
  (Total volume of hematoma and perihematomal edema on followed CT - total volume of hematoma and perihematomal edema on initial CT) / total volume of hematoma and perihematomal edema on initial CT X100%
Change in National Institutes of Health Stroke Scale (NIHSS) | Day 21±2
  NIHSS score on day 21 - initial NIHSS score. NIHSS score ranges from 0 to 42, with higher scores indicating more severe neurological deficit.
Percentage of participants with adverse events (AEs) | Day 1-21
  serious AEs (death, recurrent stroke, myocardial infarction, gastrointestinal bleeding requiring blood transfusion, etc.), nonserious AEs (abdominal pain, gastrointestinal bleeding without requiring blood transfusion, other bleeding, skin rash, etc.) Percentage of participants with serious AEs = participants with serious AEs / total participants x100% Percentage of participants with nonserious AEs = participants with nonserious AEs / total participants x100% Percentage of participants with AEs = participants with AEs / total participants x100%
modified Rankin scale (mRS) score | 3-month
  Modified Rankin scale (mRS) score is a functional outcome score, ranging from 0 to 6, with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Joe Yeh, MD PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- Natinal Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication
Access Criteria: These data will be available on the publication of this study.

REFERENCES:
- [Result] Lee SH, Park HK, Ryu WS, Lee JS, Bae HJ, Han MK, Lee YS, Kwon HM, Kim CK, Park ES, Chung JW, Jung KH, Roh JK. Effects of celecoxib on hematoma and edema volumes in primary intracerebral hemorrhage: a multicenter randomized controlled trial. Eur J Neurol. 2013 Aug;20(8):1161-9. doi: 10.1111/ene.12140. Epub 2013 Mar 29. PMID 23551657
- [Result] Dowlatshahi D, Demchuk AM, Flaherty ML, Ali M, Lyden PL, Smith EE; VISTA Collaboration. Defining hematoma expansion in intracerebral hemorrhage: relationship with patient outcomes. Neurology. 2011 Apr 5;76(14):1238-44. doi: 10.1212/WNL.0b013e3182143317. Epub 2011 Feb 23. PMID 21346218